CLINICAL TRIAL: NCT05617768
Title: Enhanced Recovery After Surgey (ERAS)Guidelines in Mitral Valve Surgeries, Questionnaire
Brief Title: Enhanced Recovery After Surgery (ERAS)Guidelines in Mitral Valve Surgeries, Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sherif Mamdouh Abbas, lecturer, Cairo University
Other Study IDs: MS-337-2022
Record Dates: First submitted 2022-10-28; First posted 2022-11-15 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: ERAS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- • Cardiac anesthesiologists • Cardiac intensivists • Cardiothoracic surgeons: * Anesthesia department, Cairo university hospitals, kasr al-ainy.
  * Cardiothoracic thoracic surgery department, Cairo university hospitals, kasr al-ainy.
  * Anesthesia department, National Heart Institute.
  * Cardiothoracic surgery department, National Heart Institute.

SUMMARY:
ERAS after cardiac surgery is a well known protocol ,However the investigators study if it is applied at our institute

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) is a term that include a series of evidence-based perioperative care pathways designed to reduce physiological and psychological stress in surgical patients and to achieve rapid recovery.

In 2016, the first pilot study was published, which analyzed enhanced recovery after cardiac surgery (ERACS). Weaning from mechanical ventilation is considered one of the items that forms the concept of enhanced recovery in cardiac surgery.

Pain is an undesirable consequence of surgery especially cardiac surgery as pain during and following cardiac surgery has been shown to be a risk factor for increased morbidity. Systemic opioids have been the main stay for the management of perioperative pain in cardiac surgery. Lower doses of opioids has been related to early extubation and minimizing opioid-related side effects, such as prolonged ventilation, tolerance, nausea, vomiting, gut dysfunction, and immunosuppression.

On the other hand the investigators find cases of morbidity and mortality not related to the surgical procedure. ERAS protocol discuss the optimum condition that can be used to avoid the morbidity and mortality complications.

the investigators aim to know how well ERAS protocol is known and applied

ELIGIBILITY:
Inclusion Criteria:

* Cardiac anesthesiologists.
* Cardiac intensivists.
* Cardiothoracic surgeons.
* All stuff members from resident to consultant are included inside this study

Exclusion Criteria:

-

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Anesthesia department, Cairo university hospitals, kasr al-ainy.
  * Cardiothoracic thoracic surgery department, Cairo university hospitals, kasr al-ainy.
  * Anesthesia department, National Heart Institute.
  * Cardiothoracic surgery department, National Heart Institute.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessement of the knowledge of doctors to ERAS guidelines in cardiac surgery by using the grading system. | 6 months
  Assessement of the knowledge of doctors to ERAS guidelines in cardiac surgery by using the grading system.Grading system will be described as:-
  * Grade A ( knows well( : more than 60 % correct answer
  * Grade B ( fair ): 35 :60 % correct answer
  * Grade C ( knows nothing ) :- less than 35 % correct answer

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Unviersity, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT05617768/Prot_SAP_001.pdf